CLINICAL TRIAL: NCT00880906
Title: Prospective, Single-Blinded, Randomized Controlled Trial With Sham Comparing Standard Therapy With or Without Esophageal Dilatation in Patients With Eosinophilic Esophagitis
Brief Title: Study of the Efficiency of Esophageal Dilation on Patient With Eosinophilic Esophagitis
Acronym: EOE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Michael Vaezi, Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 080741
Record Dates: First submitted 2008-08-25; First posted 2009-04-14 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Suspected Eosinophilic Esophagitis
Keywords: eosinophilic esophagitis; esophageal food impaction; dysphagia
MeSH Terms: conditions — Eosinophilic Esophagitis; Deglutition Disorders | interventions — Steroids; Fluticasone; Dexlansoprazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Group A receives steroids and PPI, (SOC) and esophageal dilation.
  Interventions: Procedure: Esophageal dilation; Drug: Steroid and Proton Pump Inhibitor Therapy
- B (Sham Comparator): Receives steroids and PPI only- Does not have esophageal dilation.
  Interventions: Drug: Steroid and Proton Pump Inhibitor Therapy

INTERVENTIONS:
Procedure: Esophageal dilation — The esophagus is stretched during the upper endoscopy using Maloney dilators or balloon dilatation.
  Other Names: esophageal stretching
  Arms: A
Drug: Steroid and Proton Pump Inhibitor Therapy
  Other Names: fluticasone; dexilant

SUMMARY:
This study is for patients who have had a food impaction and/or difficulty swallowing, who are scheduled to have endoscopy, biopsy and possibly dilatation (stretching) of the esophagus.

Standard treatment for people who have food impaction and difficulty swallowing is endoscopy to view the esophagus, tissue biopsies of the lining of the esophagus for diagnosis, and drug therapy including steroids and drugs used to treat reflux disease. Early dilatation or stretching of the esophagus may be done at this time but not always. Some doctors prefer to wait and see if the drugs are affective.

It is not known if dilating the esophagus early in treatment adds benefit. Therefore, we are doing this study to compare the two methods of treatment. We will compare two groups: one group will have dilatation performed during the first endoscopy and one group will not have dilatation performed during endoscopy. We will see if dilatation helps prevent food impaction and improves swallowing.

Another purpose of this study is to learn more about the causes of swallowing problems, thus extra biopsies will be taken of the esophagus and store them for future research.

DETAILED DESCRIPTION:
Eosinophilic esophagitis (EE) is an inflammatory condition of the esophagus found in the pediatric and adult population. It is characterized by an intense eosinophilic infiltration of the surface lining of the esophagus. EE is becoming an increasingly recognized diagnosis in individuals presenting with food bolus impaction and dysphagia. A history of chronic solid food dysphagia, food impaction and young age have all been noted characteristics in those patients subsequently diagnosed with EE. Eosinophilic esophagitis can be suspected by clinical presentation but histologic confirmation is necessary for a definitive diagnosis. The finding of large numbers of eosinophils (>15 per high powered field) on biopsy specimens are needed to confirm EE. Endoscopic features such as mucosal rings, linear furrows, proximal strictures and white esophageal papules have all been described in patients with EE.

The underlying pathophysiology of EE is poorly understood but is thought to be associated with a TH2-type allergic inflammatory response. Other studies have also suggested that immune dysregulation may play a role in the underlying pathophysiology of this disorder.

The optimal treatment of EE has not been determined. There have been studies noting that swallowed fluticasone propionate (FP), an inhaled corticosteroid, has shown benefit in adult and pediatric patients with EE. Esophageal dilation has been used in patients with EE with persistent dysphagia and food impaction. No study has evaluated the improvement in dysphagia and incidence of future food bolus impaction in those patients treated with early esophageal dilation. Our aim is to determine if esophageal dilation and standard drug therapy improves symptoms of dysphagia. We also plan to obtain and store esophageal biopsy specimens for future immunologic assessment to help determine the underlying pathophysiology Eosinophilic Esophagitis.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female volunteers ≥18 years old.
2. Patients with known or suspected Eosinophilic Esophagitis.
3. Patients undergoing upper endoscopy for recent food impaction or complaint of dysphagia.

Exclusion Criteria:

1. Use of oral corticosteroids.
2. Significant medical conditions that in the investigator's judgment would compromise the subject's health and safety.
3. Contraindication to esophageal dilation based on investigator's judgment.
4. Esophageal motility abnormalities not thought to be related to Eosinophilic Esophagitis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Vaezi, MD,PhD, MS epi, Principal Investigator — vanderbilt Universtiy Medical Center
Locations (1):
- Vanderbilt Unversity Medical Center Department of Gastroenterology, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A Drug Therapy Plus Dilation: Group A receives steroids and PPI, (SOC) and esophageal dilation.
  Esophageal dilation: The esophagus is stretched during the upper endoscopy using Maloney dilators or balloon dilatation.
- Group B Drug Therapy Only: Receives steroids and PPI only- Does not have esophageal dilation.
Period: Overall Study
Arm/Group | Group A Drug Therapy Plus Dilation | Group B Drug Therapy Only
Started | 29 | 21
Completed | 17 | 14
Not Completed | 12 | 7
Not completed — Lost to Follow-up | 0 | 1
Not completed — Did not meet criteria following patholog | 12 | 6

BASELINE CHARACTERISTICS:
Groups:
- Group A Receives Routine Care and Esophageal Dilatation: Group A receives steroids and PPI, (SOC) and esophageal dilation.
  Esophageal dilation: The esophagus is stretched during the upper endoscopy using Maloney dilators or balloon dilatation.
- Group B Receives SOC Only: Receives steroids and PPI only- Does not have esophageal dilation.
- Total: Total of all reporting groups
Arm/Group | Group A Receives Routine Care and Esophageal Dilatation | Group B Receives SOC Only | Total
Number analyzed (Participants) | 29 | 21 | 50
Age, Continuous [Median (Full Range); unit: Years] | 35 [19 to 61] | 32 [20 to 69] | 33 [19 to 69]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 20 | 49
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 16 | 12 | 28
Region of Enrollment [Number; unit: participants]
  United States | 29 | 21 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Dysphagia Score in Patients With Eosinophilic Esophagitis (EE)
Description: Dysphagia Scores:
  0 = able to eat normal diet / no dysphagia.
  1. = able to swallow some solid foods
  2. = able to swallow only semi solid foods
  3. = able to swallow liquids only
  4. = unable to swallow anything / total dysphagia
Time Frame: 60 days
Measure: Number; unit: Percent Change
Arm/Group | Group A Receives Routine Care and Esophageal Dilatation | Group B Receives SOC Only
Number analyzed (Participants) | 17 | 14
Percent Change | 69 | 79

2. Secondary Outcome: Immunological Assessment Into the Etiology of Eosinophilic Esophagitis
Time Frame: 60 days
Population: Saved samples were not analyzed due to there being no difference in the primary outcome measure.
Arm/Group | Group A Receives Routine Care and Esophageal Dilatation | Group B Receives SOC Only
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Group A Receives Routine Care and Esophageal Dilatation | Group B Receives SOC Only
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/14
Other Adverse Events (participants affected / at risk) | 0/17 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No